CLINICAL TRIAL: NCT06025877
Title: Quality Improvement PrecivityAD2(TM): A Survey and Clinical Utility Study of the PrecivityAD2 Blood Test in the Evaluation of Cognitive Impairment (QUIP II)
Brief Title: Quality Improvement and Clinical Utility PrecivityAD2(TM) Clinician Survey
Acronym: QUIP II
Status: Active, not recruiting | Type: Observational
Sponsor: C2N Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: C2N002
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia; Cognitive Decline; Cognitive Impairment; Memory Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Memory Disorders | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: One time clinician survey post-test following the receipt of the PrecivityAD2 blood test result
  Interventions: Other: PrecivityAD2(TM) blood test
- Cohort B: Pre-test as well as post-test and close-out survey following the receipt of the PrecivityAD2 blood test result
  Interventions: Other: PrecivityAD2(TM) blood test

INTERVENTIONS:
Other: PrecivityAD2(TM) blood test — The PrecivityAD2 blood test measures plasma amyloid beta (Aβ) peptides 42 and 40 (Aβ42/40) Ratio and phosphorylated tau (p-tau) compared to non-phosphorylated tau (np-tau) at amino acid 217 of the tau peptide (p-tau217/np-tau217) ratio to determine whether a patient with signs or symptoms of cognitive impairment is likely to have brain amyloid plaques, a pathological hallmark of AD.
  Other Names: AD2

SUMMARY:
There is a major unmet need for timely, non-invasive, and low-burden evaluation of patients presenting with mild cognitive impairment (MCI) and dementia. MCI impacts 12-18% of people in the United States over age 60 years (Alzheimer's Association. Mild Cognitive Impairment (MCI) available at https://www.alz.org/alzheimers-dementia/what-is-dementia/related_conditions/mild-cognitive-impairment. Accessed August 16, 2022). MCI does not substantially interfere with daily activities, although complex functional tasks may be performed less efficiently (Knopman DS, Petersen RC. Mild cognitive impairment and mild dementia: a clinical perspective. Mayo Clin Proc. 2014;89(10):1452-1459. doi:10.1016/j.mayocp.2014.06.019). Approximately 30% of MCI patients have Alzheimer's disease (AD) as a cause of their symptoms (Lopez,OL, Kuller LH, Becker JT, et al. Incidence of dementia in mild cognitive impairment in the cardiovascular health study cognition study. Arch Neurol. 2007;64(3):416-420.doi:10.1001/archneur.64.3.416)). In contrast, dementia is defined by chronic, acquired loss of two or more cognitive abilities caused by brain disease or injury, often associated with significant interference with the ability to function at work or at usual activities. (Knopman DS, Petersen RC. Mild cognitive impairment and mild dementia: a clinical perspective. Mayo Clin Proc. 2014;89(10):1452-1459. doi:10.1016/j.mayocp.2014.06.019). Approximately 60-80% of dementia patients have AD as a cause of their symptoms (Alzheimer's Association. Mild Cognitive Impairment (MCI) available at https://www.alz.org/alzheimers-dementia/what-is-dementia/related_conditions/mild-cognitive-impairment. Accessed August 16, 2022).

DETAILED DESCRIPTION:
The Quality Improvement PrecivityAD2(TM) Clinician Survey and Clinical Utility Study (QUIP II) represents a large-scale initiative for the PrecivityAD2 blood test for use by neurologists, geriatricians, and geropsychiatrists (memory care specialists) who see patients aged 55 years and older with signs or symptoms of MCI or dementia.

C₂N Diagnostics, LLC is a CLIA-certified, CAP-accredited diagnostic testing laboratory based in St. Louis, MO. Its new test, the PrecivityAD2 blood test, measures plasma amyloid beta (Aβ) peptides 42 and 40 (Aβ42/40) Ratio and phosphorylated tau (p-tau) compared to non-phosphorylated tau (np-tau) at amino acid 217 of the tau peptide (p-tau217/np-tau217) ratio to determine whether a patient with signs or symptoms of cognitive impairment is likely to have brain amyloid plaques, a pathological hallmark of AD.

ELIGIBILITY:
Physician Inclusion Criteria:

1. Memory care specialists actively practicing in the United States
2. Practice serves individuals with MCI or dementia age > 55 years
3. Average patient volume > 25 visits per week (all patients seen across practice)
4. Memory care specialist with access to an online electronic survey

Physician Exclusion Criteria:

1) Clinicians who practice in New York

Participant Inclusion Criteria:

1. Individual with MCI or dementia
2. Age >= 55 years

Participant Exclusion Criteria

1. Individual requiring test related blood draw within the state of New York
2. Participation does not seem to be in the best interest of the individual, per the ordering clinician

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include up to 40 memory care specialists who will use the PrecivityAD2 blood test and complete the respective surveys. Participating clinicians will be selected based on their ability to meet the acceptance measures from the inclusion and exclusion criteria. Cohort A will include up to 100 test samples collected for the PrecivityAD2 blood test. Cohort B will include up to 300 test samples collected for the PrecivityAD2 blood test.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in planned clinical management (Cohort A and B) | Day 20
  The association of the test result on medical decision making
Change in planned clinical management (Cohort B) | Day 0 vs Day 20
  Evaluate the planned versus subsequent planned change in clinical management as a result of receiving the test result
Difference between the actual age and symptomatology versus intended use criteria (Cohort A and B) | Day 90
  Evaluate the intended use criteria

SECONDARY OUTCOMES:
Relationship between the test result and actual clinical management (Cohort B) | Day 90
  Association of the test result on subsequent conducted changes in clinical management and test results when evaluating individuals with MCI or dementia in an ambulatory setting
Change in planned clinical management compared to conducted clinical management (Cohort B only) | Day 20 vs Day 90
  The evaluation of planned versus conducted change in management as a result of receiving the test result
Change in probability of AD (Cohort A and B) | Day 0 vs Day 20
  Evaluate the probability of an AD Dx pre and post receipt of the test result
Change in anti-AD medication use (Cohort A and B) | Day 0 vs Day 20
  Evaluate anti-AD medication use pre- and post-receipt of the test result
Change in diagnosis (Cohort B) | Day 0 vs Day 90
  Evaluate any changes in diagnoses as a result of receiving the AD test result
Relationship between the test result and planned testing (Cohort B) | Day 0 vs Day 20 vs Day 90
  Evaluate the association between subsequent test ordering pre and post testing
Correlations between the net promoter score and ease of use by APS2 result (Cohort B) | Day 90
  Focus group questions around net promoter score and ease of use, strengths, and limitations of testing

CONTACTS AND LOCATIONS:
Overall Officials: Mark Monane, MD, MBA, AGSF, Principal Investigator — C₂N Diagnostics, LLC
Locations (9):
- United States (9):
  - UCSF Memory and Aging Center, San Francisco, California
  - Pacific Brain Health Center, Santa Monica, California
  - Advocate Memory Center, Park Ridge, Illinois
  - Josephson Wallack Munshower Neurology, P.C., Indianapolis, Indiana
  - Tulane Doctors Neurosurgery Clinic, New Orleans, Louisiana
  - Memorial Healthcare Institute for Neuroscience, Owosso, Michigan
  - Sharlin Health and Neurology, Ozark, Missouri
  - C2N Diagnostics, St Louis, Missouri
  - Palmetto Primary Care Physicians, Summerville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monane M, Maraganore DM, Carlile RM, Johnson KG, Merrill DA, Gitelman DR, Sharlin KS, VandeVrede LA, George KK, Wang J, West T, Jacobs L, Verghese PB, Braunstein JB. Clinical Utility of an Alzheimer's Disease Blood Test Among Cognitively Impaired Patients: Results from the Quality Improvement PrecivityAD2 (QUIP II) Clinician Survey Study. Diagnostics (Basel). 2025 Jan 13;15(2):167. doi: 10.3390/diagnostics15020167. PMID 39857051